CLINICAL TRIAL: NCT03126357
Title: CSD170401: A Single-Center, Randomized, Open-Label, Crossover Study to Assess Elements of Abuse Liability for Three Electronic Tobacco Vapor Products During an 11-Day In-Clinic Confinement
Brief Title: CSD170401: Study to Assess Elements of Abuse Liability for Three Electronic Tobacco Vapor Products During an 11-Day In-Clinic Confinement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD170401
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Product usage order ABECD (Experimental): Subjects will use each of the 5 products (ABECD) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order BCADE (Experimental): Subjects will use each of the 5 products (BCADE) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order CDBEA (Experimental): Subjects will use each of the 5 products (CDBEA) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order DECAB (Experimental): Subjects will use each of the 5 products (DECAB) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order EADBC (Experimental): Subjects will use each of the 5 products (EADBC) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order DCEBA (Experimental): Subjects will use each of the 5 products (DCEBA) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order EDACB (Experimental): Subjects will use each of the 5 products (EDACB) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order AEBDC (Experimental): Subjects will use each of the 5 products (AEBDC) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order BACED (Experimental): Subjects will use each of the 5 products (BACED) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E
- Product usage order CBDAE (Experimental): Subjects will use each of the 5 products (CBDAE) sequentially for 1 and 1/2 days during an 11 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E

INTERVENTIONS:
Other: Product A — Usual Brand Cigarette
Other: Product B — FT21039 an electronic tobacco vapor product
Other: Product C — FT21092 an electronic tobacco vapor product
Other: Product D — FT21018 an electronic tobacco vapor product
Other: Product E — 4mg nicotine gum

SUMMARY:
This study will examine elements of abuse liability (AL) related to potential product adoption of three electronic tobacco vapor products by current smokers relative to high and low AL comparator products (usual brand cigarette and nicotine gum, respectively). Changes in subjective measures, speed and amount of nicotine uptake, and maximum changes in physiological effects during and after product use that follows a 12-hour (minimum) tobacco and nicotine abstinence period, will be determined. The electronic tobacco vapor products will not be compared to each other.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, crossover study, designed to evaluate subjective effects (i.e., Product Liking [PL], Overall Intent to Use Again [OIUA], Product Effects [PE], Urge to Smoke [UTS], and Overall Product Liking [OPL]), plasma nicotine uptake, and physiological measures (blood pressure and heart rate) during and following ad libitum use of the following five IPs by healthy subjects. Subjects will be evaluated in five separate Test Sessions and the active period of each Test Session will last for approximately 4 hours during and following IP use.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Able to safely perform the required study procedures, as determined by the Investigator.
4. Expired breath carbon monoxide level is ≥ 15 ppm and ≤ 100 ppm at Screening and Day 1.
5. Smokes only combustible, filtered, non-menthol cigarettes, 83 mm to 100 mm in length.
6. Agrees to smoke same usual brand (UB) cigarette throughout the study period. Usual brand cigarette is defined as the cigarette brand style currently smoked most frequently by the subject.
7. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Investigator.
8. Response at Screening to Fagerström Test for Cigarette Dependence (FTCD) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes."
9. Willing to use UB cigarette, electronic tobacco vapor products, and Nicorette gum during the study period.
10. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each Test Session.
11. Females of childbearing potential must be willing to use a form of contraception acceptable to the Investigator from the time of signing informed consent until study discharge. Examples of acceptable forms of contraception include, but are not limited to, the following.

    1. Surgeries:

       * Hysterectomy at least 6 months prior to randomization
       * Oophorectomy at least 6 months prior to randomization
       * Tubal ligation at least 6 months prior to randomization
    2. Transcervical sterilization at least 6 months prior to randomization
    3. Hormonal birth control at least 3 months prior to randomization
    4. Non-hormonal intrauterine device at least 3 months prior to randomization
    5. Double barrier methods (e.g., condom and spermicide) at least 14 days prior to randomization
    6. Abstinence at least 14 days prior to randomization
    7. Vasectomized partner is acceptable birth control for females provided the surgery was performed at least 6 months prior to randomization
    8. Postmenopausal at least 1 year prior to randomization and have follicle-stimulating hormone (FSH) levels consistent with postmenopausal status at screening as per Investigator or designee judgment
12. Agrees to in-clinic confinement of 11 days and 10 nights.

Exclusion Criteria:

1. Presence of clinically significant or unstable/uncontrolled acute or chronic medical conditions at Screening or Day 1, as determined by the Investigator, that would preclude the subject from participating safely in the study (e.g., uncontrolled hypertension, lung disease, cardiac disease, neurological disease or psychiatric disorders) based on safety assessments such as clinical laboratory tests, medical history, and physical/oral examinations.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. History or presence of stomach ulcers.
4. At risk for heart disease that would preclude the subject from participating safely in the study, as determined by the Investigator.
5. Use of medicine for the treatment of depression, unless on a stable dose for the past 6 months prior to screening and deemed clinically stable by the PI.
6. Current scheduled treatment for asthma within the past consecutive 12 months prior to screening. As needed treatment, such as inhalers, may be included at the PIs discretion pending approval from the medical monitor.
7. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
8. Systolic blood pressure of > 160 mmHg or diastolic blood pressure of > 95 mmHg at Screening, measured after being seated for at least 5 minutes.
9. Hemoglobin level is < 12 g/dL at Screening.
10. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
11. History or presence of hemophilia or any other bleeding disorders.
12. History or presence of clotting disorders and/or use of anticoagulants (e.g., clopidogrel [Plavix®], warfarin [Coumadin®, Jantoven®] and aspirin [> 325 mg/day], see Section 7.4 "Concomitant Medications").
13. Whole blood donation within 8 weeks (≤ 56 days) prior to Screening.
14. Plasma donation within (≤) 7 days prior to Screening.
15. Body mass index < 18.5 or > 40.0 kg/m2 at Screening.
16. Weight of ≤ 110 pounds at Screening.
17. Poor peripheral venous access.
18. Postponing a decision to quit smoking (defined as planning a quit attempt within [≤] 30 days of Screening) to participate in this study or previous attempt within (≤) 30 days prior to Screening.
19. Employed by a tobacco company, the study site, or handles unprocessed tobacco as part of his or her job.
20. Use of any medication or supplement that aids smoking cessation, including but not limited to any nicotine replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to Screening.
21. Use of an electronic tobacco vapor product or other tobacco or nicotine-containing product (e.g., lozenges, moist snuff) within (≤) 30 days prior to Screening.
22. Drinks more than 14 servings of alcoholic beverages per week (one serving = 12 oz of beer, 6 oz of wine, or 1.5 oz of liquor).
23. Females who have a positive pregnancy test, are pregnant, breastfeeding, or who intend to become pregnant during the course of the study.
24. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
25. A positive urine drug screen without disclosure of corresponding prescribed concomitant medication(s), at Screening or Day 1.
26. A positive alcohol result at Screening or Day 1.
27. Determined by the Investigator to be inappropriate for this study, including a subject who is unable to communicate or unwilling to cooperate with the study staff.
28. Participation in another clinical trial within (≤) 30 days prior to Screening. The 30-day window for each subject will be derived from the date of the last study event in the previous study to Screening of the current study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
AUECPL 15-240 | -5, 5, 15, 30, 45, 60, 90, 120, 150, 180, and 240 Minutes
  Area under the product liking (PL) NRS score-versus-time curve from 15 minutes to 240 minutes after the start of investigational product (IP) use.
Emax PL | -5, 5, 15, 30, 45, 60, 90, 120, 150, 180, and 240 Minutes
  Maximum response for product effects with regards to PL score after the start of IP use.
Eoverall IUA | 240 Minutes
  Overall intent to use again (IUA), measured at 240 minutes after the start of IP use.
AUCnic 0-240 | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, and 240 Minutes.
  Baseline-adjusted area under the nicotine concentration-versus-time curve from time zero to 240 minutes after the start of IP use.
Cmax | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, and 240 Minutes.
  Maximum baseline-adjusted plasma concentration.
Tmax | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, and 240 Minutes.
  Time to maximum baseline-adjusted plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tomek, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No